CLINICAL TRIAL: NCT03318796
Title: Tryton Post Approval Study (PAS) for the Tryton Side Branch Stent
Acronym: PAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tryton Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-0161
Record Dates: First submitted 2017-10-02; First posted 2017-10-24 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Coronary Artery Disease
Keywords: Bifurcation lesions
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, single arm open label registry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Interventional (Other): Coronary artery stenting of De novo bifurcation lesions MB & SB
  Interventions: Device: Coronary Artery Stenting

INTERVENTIONS:
Device: Coronary Artery Stenting — Interventional coronary artery stent placement in De novo bifurcation lesions of the MB & SB

SUMMARY:
TRYTON Post Approval Study (PAS) of the Tryton Side Branch Stent

DETAILED DESCRIPTION:
The primary objective of this PAS is to assure the continued safety and effectiveness of the Tryton Side Branch Stent™ with main branch approved DES in the treatment of de novo native coronary artery bifurcation lesions with side branch diameter ranging from ≥2.5 mm to ≤3.5 mm and main branch diameter ranging from ≥2.5 mm to ≤4.0 mm.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. The patient must be ≥18 and ≤ 90 years of age;
2. Acceptable candidate for CABG;
3. The intention to treat the side branch of the target bifurcation based on angiographic evaluation
4. The patient is willing to comply with specified follow-up evaluations;
5. The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent, approved by the appropriate Institutional Review Board (IRB).
6. Planned use of FDA approved and commercially available drug-eluting stents (DES) for subject's index procedure Angiographic Inclusion Criteria
7. a) Single de novo lesion in a bifurcation involving both the main branch and the side branch b) The bifurcation: main branch and side branch with a visual diameter stenosis ≥ 50% (Medina classification 1.1.1; 0.1.1; 1.0.1) by visual assessment;
8. Target lesion located in a native coronary artery;
9. a) Bifurcation lesion main branch reference vessel diameter must be ≥2.5 mm to ≤ 4.0 mm, and b) Side branch reference vessel diameter must be ≥2.5mm by visual estimate (≥2.25mm by QCA) and <3.5 mm by visual estimate (<3.25 mm by QCA);
10. a) Bifurcation lesion main branch lesion length ≤ 28 mm and b) Side branch lesion length ≤ 5.0 mm (the ability to be treated with a single stent for both main and side branch);
11. Target lesion ≥50% and <100% stenosed by visual estimate in both the main branch and side branch; -

Exclusion Criteria:

General Exclusion Criteria

1. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure. Female patients of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test;
2. Impaired renal function (serum creatinine >2. mg/dL or 150 μmol/l);
3. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3 or a WBC <3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis);
4. Presence of a heart transplant
5. Known allergy to cobalt chromium
6. Hypersensitivity or contraindication to cobalt-chromium or structurally-related compounds, cobalt, chromium, nickel, or tungsten
7. Anticipated use of rotational artherectomy
8. Patient in whom the use of a drug eluting stent is contraindicted, e.g., who cannot receive the recommended dual anti-platelet (aspirin and an approved P2Y12 inhibitor) and/or anticoagulant therapy

   Angiographic Exclusion Criteria:
9. Left main coronary artery disease (protected and unprotected);
10. Trifurcation lesion;
11. Totally occluded target vessels (TIMI flow 0 or 1);
12. Moderate to Severely calcified target lesion(s);
13. Highly calcified target lesion(s) requiring rotational atherectomy;
14. Target lesion has excessive tortuosity unsuitable for stent delivery and deployment;
15. Angiographic evidence of thrombus in the target lesion(s);
16. Tryton Stent placement without angioplasty pre-dilatation of the main branch and side branch (i.e., direct stenting is contraindicated)
17. Tryton Stent placement alone, without implantation of a main branch stent
18. An untreated significant (>50%) stenosis proximal or distal in either the side branch or main branch;
19. Impaired runoff in the treatment vessel with diffuse distal disease;
20. Left ventricular ejection fraction (LVEF) 30% (LVEF must be obtained within 6 months prior to the index procedure); -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 335 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) | 1 year
  Composite of cardiac death, target vessel MI (Q and non-Qwave) clinically driven target vessel revascularization

SECONDARY OUTCOMES:
Device success | 48 hrs
  Attainment of <30% residual stenosis within the side branch without device malfunction
Lesion success | 48 hrs
  Attainment of <30% residual stenosis using any percutaneous method
Procedure success | 48 hrs
  Lesion success without the occurrence of in-hospital MACE
Death | 1 year
  All-cause and cardiac mortality
Myocardial infarction (MI) | 1 year
  Q wave and Non-Q wave
CD-TLR | 1 year
  Clinically driven target lesion revascularization
CD-TVR | 1 year
  Clinically driven target vessel revascularization
Stent thrombosis | 1 year
  ARC definition of definite and probable

CONTACTS AND LOCATIONS:
Overall Officials: Joel Schnieder, MD, Principal Investigator — Rex Health; Raleigh NC
Locations (1):
- NC Heart and Vascular Research/UNC REX, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided